CLINICAL TRIAL: NCT02447926
Title: Procurement of Leukapheresis Products From End Stage Liver Disease (ESLD) Patients for Immunological Studies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Successful proof of concept study after 1 subject.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Josh Levitsky, Associate Professor of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00097231
Record Dates: First submitted 2015-04-17; First posted 2015-05-19 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: End Stage Liver Disease
Keywords: leukapheresis; regulatory T cells; liver transplantation
MeSH Terms: conditions — End Stage Liver Disease | interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Leaukapheresis of End Stage Liver Disease Patients (Other): Leukapheresis. All subjects will receive the same treatment arm.
  Interventions: Procedure: Leukapheresis

INTERVENTIONS:
Procedure: Leukapheresis — Catheter placement will occur for about 1 hour. The research nurse will schedule leukapheresis on the next day following catheter placement.
  On the day of leukapheresis, a blood draw will monitor blood counts, kidney function, liver function, and blood clotting ability. Vital signs will be checked three times over the course of intervention.
  During the procedure, blood is mixed with anticoagulant and separated (i.e. red blood cells, white blood cells, platelets, and plasma). 1-1.5 cups of white blood cells will be collected. Leukapheresis will last 3-6 hours.
  Remaining components, except for 100-200 ml of plasma, are returned through the catheter. Two teaspoons of blood will be drawn to determine when catheter removal can occur. This part of intervention lasts about 2.5-4 hours.

SUMMARY:
Regulatory CD4+CD25+ T cells (Treg) derived from the thymus and/or periphery can control immune responsiveness to auto- and allo-antigens. However, there have been few efforts to harness the therapeutic potential of isolated Tregs to control graft rejection and inducing transplantation tolerance in solid organ recipients. In order for Tregs to be used as a clinical treatment, the following properties are necessary: ex vivo generation of sufficient numbers of cells, migration in vivo to sites of antigenic reactivity, ability to suppress rejection in an alloantigen-specific manner, and survival/expansion after infusion. The and others have demonstrated 1) the feasibility of expanding Treg ex vivo, 2) the ability of these cells to down-regulate allogeneic immune responses in vitro, and 3) the efficacy of Treg for prevention of allograft rejection in animal models. In kidney transplant, the investigators have developed strategies for the ex vivo expansion of naturally occurring human Tregs (nTregs) from leukapheresis products that would allow for the clinical employment of this cellular therapy. The investigators are also interested in this approach in patients with end stage liver disease (ESLD) undergoing liver transplantation (LT). Our central hypothesis is that alloreactive human nTreg with suppressive action can be expanded ex vivo from ESLD patients (this proposal) and used to both prevent liver transplant rejection and facilitate the minimization and withdrawal of drug-based immunosuppression (future proposals). This application will further define and validate efficient methods for ex vivo expansion of human CD4+CD25+CD127- FOXP3+nTregs cells in ESLD. The investigators herein propose to use leukapheresis products obtained from patients with ESLD to further refine and optimize protocols for expansion of Tregs. Suppressive function of expanded cells will be assessed using in vitro assays of alloreactivity (mixed lymphocyte culture).

DETAILED DESCRIPTION:
Regulatory CD4+CD25+ T cells (Treg) derived from the thymus and/or periphery can control immune responsiveness to auto- and allo-antigens. However, there have been few efforts to harness the therapeutic potential of isolated Tregs to control graft rejection and inducing transplantation tolerance in solid organ recipients. In order for Tregs to be used as a clinical treatment, the following properties are necessary: ex vivo generation of sufficient numbers of cells, migration in vivo to sites of antigenic reactivity, ability to suppress rejection in an alloantigen-specific manner, and survival/expansion after infusion. We and others have demonstrated 1) the feasibility of expanding Treg ex vivo, 2) the ability of these cells to down-regulate allogeneic immune responses in vitro, and 3) the efficacy of Treg for prevention of allograft rejection in animal models. In kidney transplant, we have developed strategies for the ex vivo expansion of naturally occurring human Tregs (nTregs) from leukapheresis products that would allow for the clinical employment of this cellular therapy. We are also interested in this approach in patients with end stage liver disease (ESLD) undergoing liver transplantation (LT). Our central hypothesis is that alloreactive human nTreg with suppressive action can be expanded ex vivo from ESLD patients (this proposal) and used to both prevent liver transplant rejection and facilitate the minimization and withdrawal of drug-based immunosuppression (future proposals). This application will further define and validate efficient methods for ex vivo expansion of human CD4+CD25+CD127- FOXP3+nTregs cells in ESLD. We herein propose to use leukapheresis products obtained from patients with ESLD to further refine and optimize protocols for expansion of Tregs. Suppressive function of expanded cells will be assessed using in vitro assays of alloreactivity (mixed lymphocyte culture).

ELIGIBILITY:
Inclusion Criteria:

* >18 years old,
* ESLD MELD <25,
* No recent infection,
* no hepatic decompensation,
* no history of HIV,
* weight > 110 lbs,
* platelets > 50,000,
* HGB >10,
* no prior organ transplant

Exclusion Criteria:

* Patients ineligible for liver transplant,
* patients who do not understand why the study procedures are being conducted,
* subjects who do not meet all inclusion criteria.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Levitsky, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Comprehensive Transplant Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of the study subjects will be made from the End Stage Liver disease patients attending the outpatient pre-transplant clinics of the Northwestern Comprehensive Transplant Center.
Groups:
- Single Arm Intervention: Leukapheresis. All subjects will be assigned to the the same intervention arm.
  Leukapheresis: Catheter placement will occur for about 1 hour. The research nurse will schedule leukapheresis on the next day following catheter placement.
  On the day of leukapheresis, a blood draw will monitor blood counts, kidney function, liver function, and blood clotting ability. Vital signs will be checked three times over the course of intervention.
  During the procedure, blood is mixed with anticoagulant and separated (i.e. red blood cells, white blood cells, platelets, and plasma). 1-1.5 cups of white blood cells will be collected. Leukapheresis will last 3-6 hours.
  Remaining components, except for 100-200 ml of plasma, are returned through the catheter. Two teaspoons of blood will be drawn to determine when catheter removal can occur. This part of intervention lasts about 2.5-4 hours.
Period: Overall Study
Arm/Group | Single Arm Intervention
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Study: Leukapheresis. All subjects will receive the same treatment arm.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Regulatory CD4+CD25+ T Cells Obtained From 150 ml of Peripheral Blood in an ESLD Patient
Description: Number of regulatory CD4+CD25+ T cells after 21 days in culture from leukapheresis product (150 ml of processed blood) from ESLD patient.
Time Frame: 21 days
Measure: Number; unit: Tregs/150ml
Arm/Group | Single Arm Intervention
Number analyzed (Participants) | 1
Tregs/150ml | 10000000000

2. Primary Outcome: Suppressive Function of Expanded Cells Will be Assessed Using in Vitro Assays of Alloreactivity (Mixed Lymphocyte Culture)
Description: Assay testing - Suppressive function of expanded cells will be assessed using in vitro assays of alloreactivity (mixed lymphocyte culture). The in vitro assays will test whether the expanded Tregs will retain their suppressive function.
Time Frame: 21 days
Measure: Number; unit: percentage of Treg inhibition
Arm/Group | Single Arm Intervention
Number analyzed (Participants) | 1
percentage of Treg inhibition | 50

ADVERSE EVENTS:
Groups:
- Single Arm Treatment: Leukapheresis. All subjects will receive the same treatment arm.
  Leukapheresis: Catheter placement will occur for about 1 hour. The research nurse will schedule leukapheresis on the next day following catheter placement.
  On the day of leukapheresis, a blood draw will monitor blood counts, kidney function, liver function, and blood clotting ability. Vital signs will be checked three times over the course of intervention.
  During the procedure, blood is mixed with anticoagulant and separated (i.e. red blood cells, white blood cells, platelets, and plasma). 1-1.5 cups of white blood cells will be collected. Leukapheresis will last 3-6 hours.
  Remaining components, except for 100-200 ml of plasma, are returned through the catheter. Two teaspoons of blood will be drawn to determine when catheter removal can occur. This part of intervention lasts about 2.5-4 hours.
Arm/Group | Single Arm Treatment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
We stopped the study after one subject was enrolled because this generated enough data to support the ability to expand Tregs in our clinical laboratory to apply for a grant through the Immune Tolerance Network. Additional patients were not needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes